CLINICAL TRIAL: NCT01918501
Title: Testing Mitochondria Activity and Blood Lipid Content of Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0037-13-ZIV
Record Dates: First submitted 2013-07-02; First posted 2013-08-07 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; Remyelination; Mitochondria; fatty acids
MeSH Terms: conditions — Multiple Sclerosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood testing (Experimental): Comparison of nutrition factors in MS patients and healthy volunteers as possibly source for the pathogenesis and for the remyelination process.
  Interventions: Procedure: Blood testing

INTERVENTIONS:
Procedure: Blood testing — Blood sample will be taken once from 120 volunteers. The blood will be examine in a blind fashion, including 60 MS patients diagnosed by a neurologist based on clinical and MRI findings. The control group will include 50 age and gender match healthy volunteers and 10 more patients with unrelated neurological diseases

SUMMARY:
Background: Multiple sclerosis (MS) is a complex and multifactorial neurological disease characterized by infiltration of immune cells and progressive damage to myelin and axons. Remyelination, the generation of new myelin in the adult nervous system, is an endogenous repair mechanism that restores function of axons. Neurons require considerable energy for their activities, including synaptic neurotransmission, and hence have significant numbers of mitochondria. Unlike other cell types that are able to utilize glycolysis as an alternative energy source, glycolysis in fully differentiated neurons is basically suppressed to maintain their antioxidant status. This property makes neurons highly vulnerable to ATP deficiency, and may be a factor in the susceptibility of neurons to cell death. Mitochondria provide cellular energy by converting oxygen and nutrients into adenosine triphosphate (ATP); and reflect local metabolic needs and via oxidative phosphorylation. Nervous tissues contain about 70% lipids of their dry weight, and around 40% of these lipids are polyunsaturated fatty acids (PUFAs).

Goal: Understanding the relationship between blood composition, mitochondria role and clinical status.

Here, we will examine expression levels of different fatty acids in the blood and monitor mitochondrial transmembrane potential as marker for the mitochondria general function.

Hypothesis: Remyelination efficiency in MS is likely mediated by many factors, besides reducing inflammation. Remyelination may not be achieved correctly /sufficient in MS patients due to nutrition low content causing mitochondrial dysfunction and/or due to fatty acid molecules deficit unable to create a new myelin layer.

DETAILED DESCRIPTION:
Methods: The study will be authorized by the Ziv Helsinki Committee. Informed consent and questionnaire will obtained from all subjects before study entry. We will examine 120 volunteers in a blind fashion, including 60 MS patients diagnosed by a neurologist based on clinical, laboratory and MRI findings. Patients will be evaluated according to EDSS score. The control group will include 50 age and gender matched healthy volunteers and 10 more patients with unrelated neurological diseases. Inclusion criteria: Age 18-60; Exclusion criteria: Other diseases, pathologies, or immune system disorders. Here, we will examine expression of different fatty acids in the serum and in erythrocyte samples; Monitor mitochondrial transmembrane potential as marker for the mitochondria general function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60

Exclusion Criteria:

* Other diseases, pathologies, or immune system disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Levels of approximately 30 fatty acids in the serum and in erythrocyte samples. | Up to 2 years
  Upon enrollment, a single blood sample of approximately 20 ml will be taken. Samples of serum and in erythrocyte will be analyzed by gas chromatography mass spectrometry.

SECONDARY OUTCOMES:
Monitor mitochondrial transmembrane potential as a marker for the mitochondria general function. | Up to 2 years
  Upon enrollment, a single blood sample of approximately 20 ml will be taken. Mitochondrial transmembrane potential of platelets and lymphocytes will be analyzed by flow cytometry following specific staining.

OTHER OUTCOMES:
Develop a simple method for utilizing common flow cytometry to identify MS by examining the response of lymphocytes to myelin antigens. | Up to 2 years
  Upon enrollment, a single blood sample of approximately 20 ml will be taken. The interaction of antigen and lymphocytes induces a cascade of cellular events. We will measured responses in myelin antigen treated lymphocytes from all volunteers. After, we will utilized the fluorescence measurement of fluorescein diacetate and carboxyfluorescein diacetate succinimidyl ester (CFSE).

CONTACTS AND LOCATIONS:
Overall Officials: RADI SHAHIEN, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- ZIV Medical Center, Safed, Israel